CLINICAL TRIAL: NCT04111796
Title: Nature-based Solutions for Work-related Stress: an Intervention Study
Brief Title: Nature-based Solutions for Work-related Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Michelle Plusquin, assistant professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nature_health
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group in nature (Experimental): they participate in nature based-program during work hours
  Interventions: Other: nature based solution for stress reduction
- control group (No Intervention): they participate don't in nature based-program during work hours and perform their normal work schedule

INTERVENTIONS:
Other: nature based solution for stress reduction — participation in nature activities: 30 min stress management in nature and group activity (walking, cycling)
  Arms: group in nature

SUMMARY:
Although exposure to nature has restorative effects on human health, beneficial effects of nature-based interventions in the working environment have been underexplored. The investigators aim to conduct a randomised controlled pilot study.

During workhours one group participates in a nature-based program, the other group is a control group. The investigators test stress-related parameters including cortisol levels, wellbeing and stress, and neurocognition.

DETAILED DESCRIPTION:
Participants of the intervention group follow a 30-minute stress management course in nature followed by a nature-based activity of 1.5 hours, twice a week for 3 consecutive weeks. The investigators measure neurocognition via neurocognitive tests, emotional status via burnout assessment tool and well-being questionnaires, and asses stress levels via salivary cortisol and smartwatches.

ELIGIBILITY:
Inclusion Criteria:

* work at province of Limburg speak dutch

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognition: selective attention | 5 minutes
  computerised tests (stroop test). The scale is mean reaction time and is used as a continuous variable.
Neurocognition: short-term memory | 10 minutes
  computerised tests (Digit Span Test). The scale is number of digits and is used as a continuous variable.
Neurocognition:visual information processing speed | 5 minutes
  computerised tests (Digit Symbol test). The scale is number of digits and is used as a continuous variable.
Neurocognition: visual information processing speed | 5 minutes
  computerised tests (Pattern Comparison test ). The scale is reaction time and is used as a continuous variable.
stress levels | 5 minutes
  Assessed by salivary cortisol levels. Scale is µg/dl and used as a continuous variable.
stress levels | 10 minutes
  Assessed by questionnaires (burnout assessment tool). Scores are used as continuous variable. Lower scores represent lower risk of burnout, higher scores represent higher risk of burnout. The score is constructed from questions concerning exhaustion, mental distance, emotional disorder and cognitive disorder.
stress levels | 3 weeks
  Assessed by smartwatch (algorithm including hart rate and movement). Values are used as continuous variable

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Plusquin, Principal Investigator — Hasselt University
Locations (1):
- Province of Limburg, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No
Data will only be shared with postdoctoral researcher involved in this project in our research group. Data is pseudonymised .

REFERENCES:
- [Derived] Daniels S, Clemente DBP, Desart S, Saenen N, Sleurs H, Nawrot TS, Malina R, Plusquin M. Introducing nature at the work floor: A nature-based intervention to reduce stress and improve cognitive performance. Int J Hyg Environ Health. 2022 Mar;240:113884. doi: 10.1016/j.ijheh.2021.113884. Epub 2021 Nov 27. PMID 34847453